CLINICAL TRIAL: NCT04491435
Title: Saliva Substitute Mouthwash in NPC Survivors With Xerostomia: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FF2018-133
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Xerostomia, Hyposalivation, Saliva Substitute, Radiation-induced Toxicity, Nasopharyngeal Cancer
MeSH Terms: conditions — Xerostomia; Nasopharyngeal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessor blinded to allocation of treatment, which was only revealed after completion of data collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional (Experimental): 4 weeks use of mucin-based saliva substitute
  Interventions: Diagnostic Test: Summated Xerostomia Inventory; Diagnostic Test: Sialometry
- Control (Placebo Comparator): 4 weeks use of xylitol-based mouthwash
  Interventions: Diagnostic Test: Summated Xerostomia Inventory; Diagnostic Test: Sialometry

INTERVENTIONS:
Diagnostic Test: Summated Xerostomia Inventory — structured interview by a dedicated researcher to obtain a score of the summated xerostomia inventory (SXI)
Diagnostic Test: Sialometry — unstimulated whole saliva (UWS) flow measurement

SUMMARY:
Nasopharyngeal carcinoma (NPC) is the highest reported otorhinolaryngological malignancy reported in Malaysia affecting predominantly male adults between 40-60 years old [1, 2]. Radiation therapy (RT) has been coined as the mainstay treatment owing to its' radiosensitive properties [1, 3]. Radiation-induced DNA damage impairs proper cell division, resulting in cell death or senescence of cells that attempt to divide, particularly useful in killing malignant cells. However, radiation doses to the salivary glands cause loss of saliva producing acinar cells which ultimately hampers production of saliva in NPC patients post radiation [4]. This leads to progressive loss of salivary gland function causing xerostomia symptoms [5]. This study aims to compare the effects of two mouthwashes in the treatment of xerostomia.

DETAILED DESCRIPTION:
Xerostomia, or dry mouth caused by reduced or absent saliva flow, is a subjective symptom that can lead to impaired chewing, swallowing, altered sense of taste and speech. This eventually affects their nutritional status and quality of life. The reported prevalence of xerostomia in NPC survivors ranged from 80% -100% [6-9]. This high prevalence has stemmed a lot of interest in prevention and treatment of this important sequelae. Saliva substitute in the forms of gels, toothpaste, sprays or mouthwash has been used for treatment of xerostomia [10]. Oral7® mouthwash (Oral7 International, United Kingdom) is a mucin-based saliva substitute formulated with natural enzymes such as lactoperoxidase, lysozyme, glucose oxidase and lactoferrin, similar to naturally occuring saliva. The biophysical properties of the mouthwash can potentially provide relief to xerostomia symptoms in patients post radiotherapy translating to a better quality of life. Hence, the purpose of the present study is to evaluate the effects of saliva substitute in treating xerostomia among NPC patients post radiotherapy. The primary end-point of the study was to compare the subjective xerostomia symptoms, measured using a validated inventory taken 4 weeks following intervention and at baseline between patients who did not receive and patients who received Oral7® mouthwash. The secondary end-point was to demonstrate similar changes in objective measurements using sialometry techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed radiation therapy or concurrent chemotherapy and radiation therapy for nasopharyngeal carcinoma (clinical staging of tumour based on AJCC staging (8th edition) T1-4, N0-3, M0).
* Patients age 20 years old to 85 years old.
* Two months has elapsed since last dose of chemotherapy or radiotherapy
* Karnofsky performance score more than 70%.
* Patients complaining of xerostomia.

Exclusion Criteria:

* Those contraindicated to using mouthwash (established allergy to lactoperoxidase, lysozyme, glucose oxidase lactoferrin, cetylpyridinium chloride and xylitol)
* Patients with residual or recurrent disease.
* Patients who received intensity modulated radiation therapy.
* Patients with ongoing oral mucositis (WHO Oral Mucositis grading I to IV)
* Patients with facial, glossopharyngeal. vagus and hypoglossal nerve palsy/ paresis.
* Patients who had any form of concurrent treatment protocols (hormonal, alternative, antiviral, sialogogues or photodynamic therapy) during the study duration.
* Patients with autoimmune diseases such as systemic lupus erythematosus, rheumatoid arthritis and Sjớgren syndrome.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2020-01-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
summated xerostomia inventory (SXI) score | 4 weeks
  summated xerostomia inventory (SXI) score at baseline-summated xerostomia inventory (SXI) score at 4 weeks post intervention

SECONDARY OUTCOMES:
unstimulated whole saliva (UWS) flow | 4 weeks
  unstimulated whole saliva (UWS) flow at 4 weeks post intervention -unstimulated whole saliva (UWS) flow at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mawaddah Azman, MS, Principal Investigator — National University of Malaysia
Locations (1):
- Universiti Kebangsaan Malaysia Medical Centre, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
IPD will be shared upon publication of the research

REFERENCES:
- [Background] Gravenmade EJ, Vissink A. Mucin-containing lozenges in the treatment of intraoral problems associated with Sjogren's syndrome. A double-blind crossover study in 42 patients. Oral Surg Oral Med Oral Pathol. 1993 Apr;75(4):466-71. doi: 10.1016/0030-4220(93)90172-z. PMID 8464611
- [Derived] Marimuthu D, Han KM, Mohamad MSF, Azman M. Saliva substitute mouthwash in nasopharyngeal cancer survivors with xerostomia: a randomized controlled trial. Clin Oral Investig. 2021 May;25(5):3105-3115. doi: 10.1007/s00784-020-03634-5. Epub 2020 Nov 11. PMID 33175253